CLINICAL TRIAL: NCT02177448
Title: A Double-blind, Parallel-group Comparison Study of BIBR 277 Capsule in Patients With Essential Hypertension
Brief Title: BIBR 277 Capsule in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.267
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Enalapril

ARMS (2):
- BIBR277 and placebo matching enalapril (Experimental)
  Interventions: Drug: BIBR277 low dose; Drug: BIBR277 medium dose; Drug: BIBR277 high dose; Drug: Placebo matching enalapril
- Enalapril and placebo matching BIBR277 (Active Comparator)
  Interventions: Drug: Enalapril low dose; Drug: Enalapril medium dose; Drug: Enalapril high dose; Drug: Placebo matching BIBR277

INTERVENTIONS:
Drug: BIBR277 low dose
  Arms: BIBR277 and placebo matching enalapril
Drug: BIBR277 medium dose
  Arms: BIBR277 and placebo matching enalapril
Drug: BIBR277 high dose
  Arms: BIBR277 and placebo matching enalapril
Drug: Enalapril low dose
  Arms: Enalapril and placebo matching BIBR277
Drug: Enalapril medium dose
  Arms: Enalapril and placebo matching BIBR277
Drug: Enalapril high dose
  Arms: Enalapril and placebo matching BIBR277
Drug: Placebo matching BIBR277
  Arms: Enalapril and placebo matching BIBR277
Drug: Placebo matching enalapril
  Arms: BIBR277 and placebo matching enalapril

SUMMARY:
The efficacy and safety of Telmisartan capsule in patients with essential hypertension were evaluated in comparison with Enalapril Maleate in the double blind trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 25 years of age
* Patient is either male or female
* Outpatient. Change to inpatient is not allowed during the study period
* Blood pressure is measured 3 times or more during the 4-week observation period; the last 2 measurements in the sitting position (intervals between measurements must be less than 4 weeks) are stabilized for both of systolic pressure (within +/- 30 mmHg) and diastolic pressure within +/- 15 mmHg) with the mean exceeding 160 mmHg for systolic and 95 mmHG for diastolic pressure

Exclusion Criteria:

* Patient has severe hypertension (the last 2 measurements in the observation period exceed 120 mmHg in terms of diastolic blood pressure)
* Patient has secondary or malignant hypertension
* Patient has a history of severe cardiac failure, unstable angina, or myocardial infarction within previous six months
* Patient has atrioventricular conduction disturbance, atrial fibrillation or severe arrhythmia
* Patient has any symptoms of cerebrovascular disorder
* Patient has serious hepatic dysfunction (either GOT (glutamic-oxaloacetic transaminase) or GPT (glutamic-pyruvic transaminase) exceeds 100 U)
* Patient has renal dysfunction (serum creatinin ≥ 2.1 mg/dl)
* Patient has uncontrolled diabetic (either of the following tests exceeds the specified standards: fasting blood glucose exceeding 151 mg/dl or HbA1c exceeding 8%)
* Patient has a history of drug sensitivity to ACE (angiotensin converting enzyme) inhibitors and angiotensin II receptor antagonists
* Patient has a history of angioedema due to ACE inhibitors
* Patient has hyperkalemia (K exceeding 5.5 mEq/l)
* Patient has received enalapril just before the start of observation period
* Patient has received treatment with any other investigational drug(s) within three months of the start of observation period
* Patients is pregnant, breast-feeding, or possible pregnant, or wants to be pregnant during the study period
* Patient has any other condition that the investigator or subinvestigator feels would be inappropriate for the study participation

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 1998-09; Primary Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Antihypertensive effect | every 2 weeks up to week 12

SECONDARY OUTCOMES:
Rate of normalized blood pressure | every 2 weeks up to week 12
Occurrence of the adverse event cough | up to 12 weeks
Decrease in blood pressure (mean systolic and diastolic blood pressure) | every 2 weeks up to week 12